CLINICAL TRIAL: NCT05086120
Title: A Remote Electronically Delivered Integrated Care Pathway for Adolescents With Major Depressive Disorder: A Feasibility Study
Brief Title: A Remote Electronically Delivered Integrated Care Pathway: A Feasibility Study
Acronym: eCARIBOU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: York University (Other)
Responsible Party: Principal Investigator, Darren Courtney, Clinician Scientist with the Cundill Centre for Child and Youth Depression and a Staff Psychiatrist in the Youth Addictions and Concurrent Disorders Service, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121/2019-01
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: Tele-psychiatry; Adolescent; Depression; Measurement Based Care; Cognitive Behaviour Therapy; e-mental health
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Adolescents (age 13-18) with major depressive disorder.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Electronically Delivered Integrated Care Pathway (ICP) (Experimental): The remote electronically-delivered ICP (also known as eCARIBOU) will consist of psychiatry appointments through telemedicine every 4 weeks over 16 weeks, where the youth is at home. Prior to these appointments, measures (i.e., Mood and Feelings Questionnaire - MFQ) will be sent to the youth to be completed. Change in measure scores will be reviewed collaboratively between the psychiatrist and the youth to assist in making treatment decisions. The medication algorithm in the in-person ICP will be used to guide these decisions. The psychiatrist will also administer the Columbia Suicide Severity Rating Scale (C-SSRS) at each telepsychiatry appointment to monitor risk. Concurrently, youth will be offered internet-based Cognitive Behavioural Therapy (iCBT) and health-coaching via text.
  Interventions: Other: eCARIBOU

INTERVENTIONS:
Other: eCARIBOU — A 16 week remote electronically deliver Integrated Care Pathway (ICP) for adolescents (13-18 years old) with Major Depressive Disorder (MDD).

SUMMARY:
This is a one-armed observational study and feasibility trial of a remote electronically-delivered integrated care pathway for the treatment of adolescents. Eligible participants are between the ages of 13 and 18, inclusive, who have a primary diagnosis of major depressive disorder. Outcomes of interest are recruitment rates and participation in pathway components, including: appointments, measure-completion and use of electronically-delivered cognitive behavioural therapy.

DETAILED DESCRIPTION:
Introduction: Depression is common and debilitating in the adolescent age range. Geography or other logistical barriers may prevent youth from accessing care. Progress in the treatment of youth that uses their tendencies to engage in electronically mediated contacts (e.g., text, online videos, and livestream video chat) can strategically address depressive disorders to overcome these barriers.

Methods: The Principal Investigator will conduct a pilot single-arm trial to assess the feasibility of a 16-week remote electronically delivered integrated care pathway (ICP) for the treatment of adolescents (age 13-18) with major depressive disorder. CBT components being delivered has been tested in the age 18-30 with depression. The ICP includes: tele-psychiatry appointments, online measurement-based care, internet-based cognitive behavioural therapy combined with mindfulness training, and text-based health coaching. Eligible subjects will be recruited from Child, Youth and Family services at the Centre for Addiction and Mental Health. The Principal Investigator aims to recruit 12 participants.

Outcomes: Feasibility outcomes are of the primary interest; namely, recruitment rates, proportion of psychiatry appointments attended, proportion of self-report measures completed, proportion of online CBT videos viewed, number of text-exchanges between youth and health coaches, physical activity levels and qualitative feedback from youth about their experiences. Primary clinical outcomes will be described via self-reported depressive symptoms using the Mood and Feelings Questionnaire. Secondary outcomes include self-reported anxiety (anxiety-related subscales of the Revised Children's Anxiety and Depression Scale) and function (Youth Columbia Impairment Scale). The Principal Investigator will also measure self-injurious thoughts and behaviours using the Columbia Suicide Severity Rating Scale.

Discussion: If results confirm hypotheses that youth can be feasibly treated with a remote electronically delivered ICP, further efficacy testing may be performed to assess this as a viable option for service delivery that reduces barriers to care.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years old at baseline
* Mood and Feelings Questionnaire - Childhood, long version (MFQ) score of ≥22
* Diagnosis of Major Depressive Disorder by impression from the referring psychiatrist and confirmed using the KSADS
* Internet access at home
* Access to a smartphone for personal and private use, with an associated standard data plan (ie. greater than or equal to 500 MB/month)
* Able to speak and read English fluently

Exclusion Criteria:

* Individuals that arecurrently receiving structured psychotherapy
* Clinically significant suicidal ideation that is defined as 'imminent intent' or attempted suicide in the past 6 months
* Co-morbid diagnosis of borderline personality disorder (as assessed by the Childhood Interview for Borderline Personality Disorder) (Zanarini, 2003), schizophrenia, bipolar disorder, moderate-to-severe eating disorder, obsessive compulsive disorder and/or severe alcohol/substance use disorder in the past 3 months
* Youth with known or clinically suspected intellectual disability or autism spectrum disorder
* Youth who are not able to provide informed consent for any other reason

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Recruitment | 6 months
  Time it takes to recruit 12 participants to the study
Number of Psychiatry Appointments | 16 weeks
  Proportion of scheduled psychiatry appointments attended (number attended divided by 4 for each participant)
Number of iCBT Content Viewed | 16 weeks
  Proportion of online CBT videos viewed per participant (number viewed divided by 54)
Number of Health Coach Text Messages | 16 weeks
  Number of text messages the participant sent to the health coach (count data)
Fitbit Usage | 16 weeks
  Number of days the fitbit is worn and the percentage of data collected
Psychiatric Management | 16 weeks
  Number of events involving of self-harm behaviour/suicidal ideation that required acute psychiatric management (where the study psychiatrist needs to communicate with the youth and/or family members outside of regular appointments every 4 weeks).
Youth's Experience with eCARIBOU | 16 weeks
  Qualitative Interview feedback from youth pertaining to the intervention - including ease of use, content relevance, level of engagement with the intervention
ICP Deviations | 16 weeks
  Frequency of deviations from the pathway and any documented reasons for deviations

CONTACTS AND LOCATIONS:
Overall Officials: Darren Courtney, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - The Center for Addiction and Mental Health, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ritvo P, Knyahnytska Y, Pirbaglou M, Wang W, Tomlinson G, Zhao H, Linklater R, Bai S, Kirk M, Katz J, Harber L, Daskalakis Z. Online Mindfulness-Based Cognitive Behavioral Therapy Intervention for Youth With Major Depressive Disorders: Randomized Controlled Trial. J Med Internet Res. 2021 Mar 10;23(3):e24380. doi: 10.2196/24380. PMID 33688840